CLINICAL TRIAL: NCT01469962
Title: Evolution of Fibrosis Scores During Weight Loss in a Population of Patients Operated on for Morbid Obesity
Brief Title: Evaluation of Liver Fibrosis Following Surgical-induced Weight Loss
Acronym: FIBROTEST
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Collaborators: University Hospital, Lille (Other); Amiens University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/079/HP
Record Dates: First submitted 2011-11-05; First posted 2011-11-10 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Obesity
Keywords: morbid obesity; bariatric surgery; NASH; Liver fibrosis; Fibrotest
MeSH Terms: conditions — Obesity; Obesity, Morbid; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- obese patients

SUMMARY:
Obesity is a frequent disease with an increased prevalence, estimated to 12.4% in France (OBEPI study 2006). Non alcoholic fatty liver disease (NAFLD) and non alcoholic steatohepatitis (NASH) both complicate morbid obesity and could be responsible for the development of liver fibrosis and consequently of liver cirrhosis. Bariatric surgery has been widely used in obese patients to reduce their weight but also to decrease morbidity conditions related to obesity. It could be involved in an improvement in liver lesions observed in obese patients. To evaluate the severity of liver lesions, the gold standard is pathological examination of the liver using percutaneous or surgical biopsies, with a scoring called Fibrosis score stage. Alternative less invasive techniques have been developed to evaluate liver lesions. These tests are commonly used in clinical hepatology and consisted of serum levels determination of fibrosis markers (Fibrotest, Transthyretin).

The aim of this study is to evaluate the evolution of fibrosis scores during weight loss in a population of patients operated on for morbid obesity ( BMI > 40kg/m2 or BMI> 35kg/m2 with comorbidity). The primary end point is to evaluate the concordance between Fibrotest and transthyretin serum levels. The number of patients has been calculated on the basis of a concordance ( Kendall test) superior to 70% in patients with grade F1 fibrosis that represents about 40% of morbid obese patients. A total of 255 patients has to be enrolled in this study. According to the number of patients operated on in the 3 centres (>150/year), the time for recruitment is 12 months. Secondary end points will evaluate in these patients the excess weight loss, the improvement in fibrosis liver tests and the correlation with improvement in other obesity- related conditions, according to surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* patients operated on for morbid obesity (BMI >40kg/m2 or >35kg/m2 associated with comorbidity)

Exclusion Criteria:

* contraindications to morbid obesity surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: obese patients
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2011-11; Primary Completion 2013-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Improvement in transthyretin serum levels | 1 year after surgery
  We will measure the modifications of Transthyretin serum levels in correlation with fibrotest, one year after surgery, to assess the effect of weight loss on liver fibrosis

SECONDARY OUTCOMES:
improvement in fibrosis scores (fibrotest, nashtest, steatotest) | 1 year after surgery
  We will measure the modifications of fibrosis scores, one year after surgery, to assess the effect of weight loss on liver fibrosis

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France